CLINICAL TRIAL: NCT04014036
Title: Treatment of Chronic Prostatitis/ Pelvic Pain Syndrome With Low-intensity Extracorporeal Shockwave Therapy: A Prospective, Randomized, Single-blind, Cross-over Study
Brief Title: Treatment of Chronic Prostatitis/ Pelvic Pain Syndrome With Low-intensity Extracorporeal Shockwave Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University (Other)
Responsible Party: Principal Investigator, Fu-Shun Hsu, Principal Investigator, National Taiwan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NTUH-57401-19
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Chronic Prostatitis/ Pelvic Pain Syndrome
Keywords: chronic prostatitis/ pelvic pain syndrome; low-intensity extracorporeal shockwave therapy

STUDY DESIGN:
Intervention Model Description: We prospectively assessed the clinical outcome of LI-ESWT for the treatment of CPPS. This study was approved by the institutional review board at National Taiwan University Hospital (NTUH, No. T-NTUH-57401).
Who Masked: Participant
Masking Description: While subjects receive Sham therapy, the machine turning on but the energy is zero.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): 30 subjects receive ESWT (LM-IASO, Litemed Co., Taiwan) for 6 courses in 3 weeks (0.05mJ/mm2, 3000 pulses). Thereafter, the two groups are cross over.
  Interventions: Device: low energy extracorporeal shockwave therapy
- 2 (Sham Comparator): 30 subjects receive Sham therapy for 3 weeks (the machine turning on but the energy is zero). Thereafter, the two groups are cross over.
  Interventions: Device: low energy extracorporeal shockwave therapy

INTERVENTIONS:
Device: low energy extracorporeal shockwave therapy — Low-intensity extracorporeal shockwave therapy (LI-ESWT) was proved to be useful in various medical conditions; for example, neovascularization in myocardial ischemia, nonhealing wounds, ED and chronic pelvic pain syndrome

SUMMARY:
This study is a prospective, randomized, single-blinded, cross-over trial to investigate the efficacy of low-intensity extracorporeal shockwave therapy in the treatment of chronic pelvic pain syndrome (CPPS). We will enroll 60 subjects with Chronic Prostatitis Symptom Index (CPSI) > 15. 30 subjects receive ESWT (LM-IASO, Litemed Co., Taiwan) for 6 courses in 3 weeks (0.05mJ/mm2, 3000 pulses) and 30 subjects receive Sham therapy for 3 weeks (the machine turning on but the energy is zero). After 3 weeks, the two groups are cross over, for additional 6 courses. The primary outcome is the the 4th week change from baseline for CPSI score. Secondary outcomes are the 8th week change from baseline for CPSI score, IIEF, QoL; AEs. The between-group relationships of baseline and 4-week data were evaluated by using the Student's t-test or Mann-Whitney U-test where appropriate. Multiple linear regression was carried out to test the variables associated with treatment outcome. P-values < 0.05 were considered statistically significant.

DETAILED DESCRIPTION:
Low-intensity extracorporeal shockwave therapy (LI-ESWT) was proved to be useful in various medical conditions; for example, neovascularization in myocardial ischemia, nonhealing wounds, ED and chronic pelvic pain syndrome.

The use of LI-ESWT has been increasingly proposed as a treatment for CPPS over the last decade. Overall, most of these studies reported encouraging results, regardless of variation in LI-ESWT set-up parameters or treatment protocols. As a whole these studies suggest that LI-ESWT could significantly improve the CPSI score and pain symptoms of CPPS patients. However, no randomized control trial with cross-over designed studies so far.

This is a prospective, randomized, single-blind, cross-over clinical study. This study will be performed in outpatient setting of NTUH. Written informed consent will be given by all participants before entering the study. The subjects are treated at the therapy room of the department of urology, NTUH. All subjects would not pay any cost for this treatment/study. This study was approved by the institutional review board at National Taiwan University Hospital (NTUH, No. T-NTUH-57401).

Inclusion criteria: were patient age 20 ~ 70 year-old man, suffering from CPPS for over 3 months, and CPSI >15. The written informed consent forms from all subjects who met the inclusion criteria were obtained.

Exclusion criteria: Patients with penile implant, prior radical prostatectomy, rectal surgery, radiation therapy to the pelvic area, spinal cord injury, prostate cancer, bladder cancer, interstitial cystitis, or major depression were excluded.

Measurement of outcomes

Primary outcome: the 4th week and the 8th week change from baseline for CPSI score.

Secondary outcomes: International Index of Erectile Function Questionnaires (IIEF) at 4th and 8th week, QoL; AEs

Methodology: All patients diagnosed of CPPS will be treated at out-patient clinic. 30 subjects receive LI-ESWT (LM-IASO, Litemed Co., Taiwan) for 6 courses in 3 weeks (0.05mJ/mm2, 3000 pulses) and 30 subjects receive Sham therapy for 3 weeks (the machine turning on but the energy is zero). LI-ESWT is delivered by a probe that was attached to a electrohydraulic unit with a wide-focused shockwave source. The shockwaves are delivered at perineum area. The duration of each ESWT session is about 20 minutes, and comprised 3000 pulses (0.05mJ/mm2), and a frequency of 100/min. After 3 weeks, the two groups are cross over.

Safety Considerations The peri- and post-treatment adverse events (AEs), including local pain, edema or hematoma were recorded and compared. With consideration of safety issue, any moderate/severe local pain or hematoma would be immediately reported and well inspected.

Follow-up The following parameters are assessed before treatment and weekly during the treatment: CPSI score, IIEF, QoL; AEs.

ELIGIBILITY:
Inclusion Criteria:

Suffering from CPPS over 3 months CPSI >15

Exclusion Criteria:

1. Patient with prior radical prostatectomy, rectal surgery, radiation therapy to the pelvic area, spinal cord injury, prostate cancer, bladder cancer, or known interstitial cystitis.
2. Have major depression or any major psychogenic disorders.
3. Patients with penile implant.

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
CPSI score | the 4th week and the 8th week
  the 4th and the 8th week change from baseline for CPSI score.
  1. In the last week, have you experienced any pain / discomfort?
     1. perineum
     2. Testicles
     3. Tip of the penis
     4. pubic area
  2. In the last week, have you:
     1. Pain or burning during urination?
     2. discomfort after sexual climax?
  3. How often have you had pain over the last week? 0 Never ~ 5 Always
  4. Which number describes your AVERAGE pain / discomfort over the last week? 0 ~10
  5. How often have you had a sensation of not emptying your bladder completely after you finished urinating? 0 Not at all ~ 5 Almost always
  6. How often have you had to urinate again <2 hours you finished urinating? 0 Not at all ~ 5 Almost always
  7. Your symptoms kept you over the last week? 0 None ~ 3 A lot
  8. How much did you think about your symptoms, over the last week? 0 None ~ 3 A lot
  9. If your symptoms persists during the rest of your life, how would how would you feel? 0-6

SECONDARY OUTCOMES:
IIEF-5 score | the 4th week and the 8th week
  Over the past 6 months:
  How do you rate your confidence that you could get and keep an erection? (1-5) When you had erections with sexual stimulation, how often were your erections hard enough for penetration? (1-5) During sexual intercourse, how often were you able to maintain your erection after you had penetrated your partner? (1-5) During sexual intercourse, how difficult was it to maintain your erection to completion of intercourse? (1-5) When you attempted sexual intercourse, how often was it satisfactory for you? (1-5) Total Score: 1-7: Severe ED 8-11: Moderate ED 12-16: Mild-moderate ED 17-21: Mild ED 22-25: No ED

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Shun Hsu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sokolakis I, Hatzichristodoulou G. Clinical studies on low intensity extracorporeal shockwave therapy for erectile dysfunction: a systematic review and meta-analysis of randomised controlled trials. Int J Impot Res. 2019 May;31(3):177-194. doi: 10.1038/s41443-019-0117-z. Epub 2019 Jan 21. PMID 30664671
- [Background] Campbell JD, Trock BJ, Oppenheim AR, Anusionwu I, Gor RA, Burnett AL. Meta-analysis of randomized controlled trials that assess the efficacy of low-intensity shockwave therapy for the treatment of erectile dysfunction. Ther Adv Urol. 2019 Mar 29;11:1756287219838364. doi: 10.1177/1756287219838364. eCollection 2019 Jan-Dec. PMID 30956690
- [Background] Dong L, Chang D, Zhang X, Li J, Yang F, Tan K, Yang Y, Yong S, Yu X. Effect of Low-Intensity Extracorporeal Shock Wave on the Treatment of Erectile Dysfunction: A Systematic Review and Meta-Analysis. Am J Mens Health. 2019 Mar-Apr;13(2):1557988319846749. doi: 10.1177/1557988319846749. PMID 31027441